CLINICAL TRIAL: NCT00854529
Title: Subconjunctival Bevacizumab Injection for the Prevention of Bleb Vascularization Post Trabeculectomy
Brief Title: Subconjunctival Bevacizumab Effect on Bleb Vascularity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Moshe Lusky / MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 005285
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Bleb Vascularity; Bleb Fibrosis; Trabeculectomy Failure
Keywords: bevacizumab; subconjunctival injection; trabeculectomy; bleb; mitomycin c
MeSH Terms: conditions — Blister | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 20 patients who had an uneventful trabeculectomy with usage of mitomycin C, will receive subconjunctival bevacizumab 1 week after the surgery
  Interventions: Drug: Bevacizumab
- 2 (Active Comparator): 20 patients who had an uneventful trabeculectomy with usage of mitomycin C, will receive subconjunctival bevacizumab 2 weeks after the surgery
  Interventions: Drug: Bevacizumab
- 3 (No Intervention): 20 patients after an uneventful trabeculectomy with usage of mitomycin C, will not receive any bevacizumab injection.

INTERVENTIONS:
Drug: Bevacizumab — sub-conjunctival injection of 1.25mg Bevacizumab
  Other Names: Avastin
  Arms: 1; 2

SUMMARY:
Trabeculectomy is an ocular surgery intended to reduce intra-ocular pressure the surgery creates a sub-conjunctival filtering bleb which filters aqueous humor fluid out.

A rather common adverse event of the surgery is increasing vascularity of the conjunctiva overlying the bleb. This leads to adherence of the conjunctiva to the sclera and fibrosis and finally failure of the bleb (and of the surgery) this study intends to demonstrate that post operative subconjunctival bevacizumab injection will reduce incidence of bleb vascularity and ultimately, bleb failure.

DETAILED DESCRIPTION:
trabeculectomy is an ocular surgery intended to reduce intra-ocular pressure the surgery creates a sub-conjunctival filtering bleb which filters aqueous humor fluid out.

a rather common adverse event of the surgery is increasing vascularity of the conjunctiva overlying the bleb. this leads to adherence of the conjunctiva to the sclera and fibrosis and finally failure of the bleb (and of the surgery) this study wishes to demonstrate that post operative subconjunctival bevacizumab injection will reduce incidence of bleb vascularity and ultimately, bleb failure.

during the study, one study group will be given subconjunctival bevacizumab 1 week after surgery, another study group will be given subconjunctival bevacizumab 2 week after surgery, and a third group will serve as control and will not receive bevacizumab. if bleb vascularity will be diagnosed all patients will be treated according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* post uneventful trabeculectomy with mitomycin c application during surgery
* adult

Exclusion Criteria:

* usage of 5-fluorouracil in trabeculectomy
* post-operative complications
* ischemic heart disease
* s/p cerebrovascular accident
* allergy to bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Bleb vascularity grading | 1, 2, 3, 4, 5. 6. montes post operative.

SECONDARY OUTCOMES:
Indiana Bleb Appearance Grading Scale (IBAGS) | 1, 2, 3, 4, 5, 6 months post operative
Intra-ocular pressure | 1, 2, 3, 4, 5, 6 months post operative
Indication for subconjunctival Mitomycin C injection or revision of surgery = yes / no | 1, 2, 3, 4, 5, 6 months post operative

CONTACTS AND LOCATIONS:
Overall Officials: moshe lusky, MD, Principal Investigator — Rabin Medical Center; omer Y bialer, MD, Study Chair — rabin medial center; anat robinson, MD, Study Chair — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Ichhpujani P, Ramasubramanian A, Kaushik S, Pandav SS. Bevacizumab in glaucoma: a review. Can J Ophthalmol. 2007 Dec;42(6):812-5. doi: 10.3129/i07-160. PMID 18026201
- [Result] Schwartz AL, Van Veldhuisen PC, Gaasterland DE, Ederer F, Sullivan EK, Cyrlin MN. The Advanced Glaucoma Intervention Study (AGIS): 5. Encapsulated bleb after initial trabeculectomy. Am J Ophthalmol. 1999 Jan;127(1):8-19. doi: 10.1016/s0002-9394(98)00290-6. PMID 9932993
- [Result] Grewal DS, Jain R, Kumar H, Grewal SP. Evaluation of subconjunctival bevacizumab as an adjunct to trabeculectomy a pilot study. Ophthalmology. 2008 Dec;115(12):2141-2145.e2. doi: 10.1016/j.ophtha.2008.06.009. Epub 2008 Aug 9. PMID 18692246
- [Result] Coote MA, Ruddle JB, Qin Q, Crowston JG. Vascular changes after intra-bleb injection of bevacizumab. J Glaucoma. 2008 Oct-Nov;17(7):517-8. doi: 10.1097/IJG.0b013e31815f5345. PMID 18854726
- [Result] Kahook MY, Schuman JS, Noecker RJ. Needle bleb revision of encapsulated filtering bleb with bevacizumab. Ophthalmic Surg Lasers Imaging. 2006 Mar-Apr;37(2):148-50. PMID 16583638
- [Result] Treatment of Failing Blebs with Ranibizumab. Study number NCT00570726. http://clinicaltrials.gov